CLINICAL TRIAL: NCT04301843
Title: Phase II Trial of Eflornithine (DFMO) and Etoposide for Relapsed/Refractory Neuroblastoma
Brief Title: Eflornithine (DFMO) and Etoposide for Relapsed/Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: K C Pharmaceuticals Inc. (Industry); Beat NB Cancer Foundation (Other); Team Parker for Life (Unknown); USWM, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Chair, Beat Childhood Cancer, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC015
Expanded Access: NCT03581240 (Available)
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eflornithine (DFMO) (Experimental): In this study subjects will receive six 21-day cycles of Etoposide and DFMO followed by an additional 630 days of DFMO alone.
  Etoposide will be given at 50 mg/m2/dose PO daily for the first 14 days of each 21 days until 6 cycles of etoposide are completed.
  DFMO (difluoromethylornithine) will be given at a dose of 1000 mg/m2 BID on each day of study.
  Interventions: Drug: Eflornithine

INTERVENTIONS:
Drug: Eflornithine — DFMO (difluoromethylornithine) will be given at a dose of 1000 mg/m2 BID on each day of study.
  Other Names: DFMO; difluoromethylornithine

SUMMARY:
Difluoromethylornithine (DFMO) will be used in an open label, multicenter, study in combination with etoposide for subjects with relapsed/refractory neuroblastoma.

DETAILED DESCRIPTION:
Difluoromethylornithine (DFMO) will be used in an open label, multicenter, study in combination with etoposide for subjects with relapsed/refractory neuroblastoma.

In this study subjects will receive six 21-day cycles of Etoposide and DFMO followed by an additional 630 days of DFMO alone.

Subjects will be evaluated in 3 arms:

• Arm 1: Subjects who show no active disease after receiving any additional therapy for neuroblastoma that was refractory to standard induction/consolidation therapy.

Refractory: Subjects with progressive disease on upfront therapy OR did not have at least PR on induction OR required additional second line therapy to achieve remission who are now in first remission.

* Arm 2: Subjects who have previously relapsed and currently show no active disease (in CR2 or greater).
* Arm 3: Subjects who are relapsed or refractory with active disease.- CLOSED TO ENROLLMENT

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a pathologically confirmed diagnosis of neuroblastoma, ≤ 30.99 years of age with history of relapsed/refractory neuroblastoma.
* All patients must have completed upfront therapy with at least 4 cycles of aggressive multi-drug chemotherapy.
* Specific Criteria by Arm:

Arms 1 and 2:

Subjects with no active disease:

i. No evidence of residual disease by CT/MRI and MIBG scan (or PET for patients who have a history of MIBG non-avid disease).

o Note: Patients with residual masses detected by CT/MRI may be considered in CR if their MIBG is negative or if MIBG positive and evaluated by PET and found to have negative PET scans; biopsy confirmation may be considered if there is still reasonable concern for persistent disease but is not required.

ii. No evidence of disease metastatic to bone marrow.

Arm 3 [CLOSED TO ENROLLMENT]:

Measurable or evaluable disease, including at least one of the following:

Measurable tumor by CT or MRI; or a positive MIBG and PET; or positive bone marrow biopsy/aspirate in at least one site.

* Timing from prior therapy: Enrollment (first dose of DFMO) no later than 60 days from last dose of the most recent therapy.
* Subjects must have fully recovered from the acute toxic effects of all prior anti- cancer chemotherapy and be within the following timelines:

  1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
  2. Hematopoietic growth factors: At least 5 days since the completion of therapy with a growth factor.
  3. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
  4. Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines, CAR-T cells.
  5. Anti-GD2 Monoclonal antibodies: At least 2 weeks must have elapsed since prior treatment with a monoclonal antibody.
  6. XRT: At least 14 days since the last treatment except for radiation delivered with palliative intent to a non-target site.
  7. Stem Cell Transplant:

     1. Allogeneic: No evidence of active graft vs. host disease
     2. Allo/Auto: ≥ 2 months must have elapsed since transplant.
  8. MIBG Therapy: At least 8 weeks since treatment with MIBG therapy
* Subjects must have a Lansky or Karnofsky Performance Scale score of 60% or higher.
* Life expectancy > 2 months
* All clinical and laboratory studies for organ functions to determine eligibility must be performed within 7 days prior to first dose of study drug unless otherwise indicated below.
* Subjects must have adequate organ functions at the time of registration:

  * Hematological: Total absolute neutrophil count ANC ≥750/μL
  * Liver: Subjects must have adequate liver function as defined by AST and ALT <5x upper limit of normal (Normal=45), Bilirubin <1.5x upper limit normal (Normal=1.0). Normal PT, PTT, fibrinogen.
  * Renal: Estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70.

The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr

* Subjects of childbearing potential must have a negative pregnancy test. Subjects of childbearing potential must agree to use an effective birth control method. Subjects who are lactating must agree to stop breast-feeding.
* Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or patients' legal representative).

Exclusion Criteria:

* BSA of <0.25 m2.
* Subjects that received DFMO at a dose higher than 1000mg/m2 BID prior to this study are not eligible.
* Subjects that received a dose of DFMO in combination with etoposide are not eligible.
* Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from hematological and bone marrow suppression effects of prior chemotherapy.
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with event free survival (EFS) during study | 2 years plus 5 years follow up
  To evaluate the efficacy of difluoromethylornithine (DFMO) in combination with etoposide in patients with relapsed/refractory neuroblastoma, based upon:
  o Event free survival (EFS) from time of enrollment.

SECONDARY OUTCOMES:
Length of time that participants experience Overall Survival (OS) | 7 years
  To evaluate the efficacy of difluoromethylornithine (DFMO) in combination with etoposide in patients with relapsed/refractory neuroblastoma, based upon:
  o Overall Survival (OS) from time of enrollment.
Determine the Overall Response Rate (ORR) of Participants using INSS Response Evaluation Criteria. | 2 years
  To evaluate the efficacy of difluoromethylornithine (DFMO) in combination with etoposide in patients with relapsed/refractory neuroblastoma, based upon:
  o Response Rate for patients with active disease (Arm 3) using International Neuroblastoma Staging System (INSS) Response Evaluation Criteria.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To monitor the safety and tolerability profile of difluoromethylornithine (DFMO) in combination with etoposide in pediatric and young adult patients with relapsed/refractory neuroblastoma.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer
Locations (31):
- United States (25):
  - University of Alabama/Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Augusta University Health, Augusta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - UHC Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CHUQ, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — https://research.beatcc.org/